CLINICAL TRIAL: NCT04090671
Title: Das Multidimensionale Dyspnoe Profil (MDP) Bei COPD, Herzinsuffizienz Und Schlafapnoe
Brief Title: Evaluation of the Multidimensional Dyspnea Profile (MDP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut für Pneumologie Hagen Ambrock eV (Industry)
Responsible Party: Principal Investigator, Georg Nilius, Prof DR med, Prof. Dr. med., Kliniken Essen-Mitte
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MDP2018
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: COPD Exacerbation; CHF; OSA; COPD
Keywords: Dyspnoea; MDP
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Intervention Model Description: multicenter prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- COPD Exacerbation (Active Comparator): the questionnaire MDP will be administered at the day of hospital admission and at the day of discharge.
  Interventions: Diagnostic Test: Multidimensional Dyspnea Profile
- CHF (Active Comparator): the questionnaire MDP will be administered at the day of hospital admission and at the day of discharge.
  Interventions: Diagnostic Test: Multidimensional Dyspnea Profile
- COPD (Active Comparator): In stable state of COPD, the questionnaire MDP will be administered once during a routine control visit at the hospital or the medical practice.
  Interventions: Diagnostic Test: Multidimensional Dyspnea Profile
- OSA (Active Comparator): The questionnaire MDP will be administered once during the first visit in the sleep laboratory.
  Interventions: Diagnostic Test: Multidimensional Dyspnea Profile

INTERVENTIONS:
Diagnostic Test: Multidimensional Dyspnea Profile — The Multidimensional Dyspnea Profile measures the intensity of dyspneic breathing discomforts. It tests five sensory qualities that describe the patient's dyspnea in its respective intensity. Additionally it includes five potential reactions. The MDP is designed to refer to a specific event of time.
  Other Names: MDP

SUMMARY:
Aim of this multicenter prospective cohort study is the evaluation of the multidimensional qualities of dyspnea in a number of diseases using the Multidimensional Dyspnea Profile (Banzett et al, ERJ 2015).

DETAILED DESCRIPTION:
The study sites will examine patients with COPD (Chronic obstructive pulmonary disease) in state of acute exacerbation and in stable state, patients with congestive heart failure (CHF) in state of acute decompensated cardiac insufficiency, and patients newly diagnosed with obstructive sleep apnea (OSA) as a control group.

In the acute setting of COPD and CHF, the questionnaire will be given at the day of hospital admission and at the day of discharge. The patients will additionally fill the Severe Respiratory Insufficiency (SRI) Questionnaire (in COPD) or the Physical Activity Questionnaire 50+ (in CHF).

In stable state of COPD, the questionnaires will be given once during a routine control visit at the hospital or the medical practice.

In OSA, the questionnaire will be given once during the first visit in the sleep laboratory.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients with acute exacerbation (Group I)
* CHF patients with acute decompensation (group II)
* stable COPD patients (group III)
* OSA patients with AHI>15 (group IV)

Exclusion Criteria:

* Other severe acute diseases that contradict the participation in a clinical trial
* Simultaneous participation in another clinical trial
* Not capable of giving consent
* Language abilities and other disabilities that contradicts the understanding or completing of a clinical questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-12-19 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
MDP scores during hospital stay | day 1 to day 5
  A1, Scale: Scale about breathing sensations with a defined start- and endpoint (neutral - unbearable). Values reach from 0-10, and higher values represent a worse outcome.
  SQ1 (sensoric quality), Choice: 5 Phrases and terms about breathing sensations. Choose between yes and no and select one as "most accurately".
  SQ2 (sensoric quality), Scales: 5 subscales about intensity of breathing sensations (muscle work; air hunger; chest tightness; mental effort; breathing a lot) with defined start- and endpoints (none - as intense as imaginable). Values reach from 0 - 10, and higher values represent a worse outcome.
  A2 (emotional quality), Scales: 5 subscales about emotions (depressed, anxious, frustrated, angry, afraid) with defined start- and endpoints (none - as intense as imaginable). Values reach from 0 - 10, and higher values represent a worse outcome.

SECONDARY OUTCOMES:
comparison of MDP scores with clinical data | 1 to 5 (+- 3) days
  comparison of the A1 and A2 (scale 0-10) and SQ2 (scale 0-10) scores of the MDP between the diseases, the evaluation of dependencies of clinical routine data with the MDP scores

CONTACTS AND LOCATIONS:
Overall Officials: Georg Nilius, Prof.Dr.med, Principal Investigator — KEM Kliniken Essen-Mitte
Locations (4):
- Germany (4):
  - Kliniken Essen-Mitte, Evang. Huyssens-Stiftung/Knappschaft gGmbH, Essen, North Rhine-Westphalia
  - Helios Klinik Hagen Ambrock, Hagen, North Rhine-Westphalia
  - Märkische Kliniken GmbH, Klinikum Lüdenscheid, Lüdenscheid, North Rhine-Westphalia
  - Praxis Dr. med V. Jansen, Menden, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No